CLINICAL TRIAL: NCT04671212
Title: Discarded Bone Marrow for Hematology Research
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BMHR
Record Dates: First submitted 2020-12-02; First posted 2020-12-17 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hemoglobinopathies
Keywords: Bone samples; Bone marrow; Discarded; Hemoglobinopathies; Non-hemoglobinopathies
MeSH Terms: conditions — Hemoglobinopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow-containing bone samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthopedic Surgery Patients: Participants receiving orthopedic surgery for clinical management that involve bone marrow containing bone discard.

SUMMARY:
The primary objective of this study is to establish a mechanism to obtain discarded bone marrow-containing bone samples from hemoglobinopathy, as well as non-hemoglobinopathy individuals. The processing of samples will help to understand how best to manipulate HSPC's from hemoglobinopathy patients with gene therapy and gene technologies in the laboratory environment. It will also allow us to establish a reservoir of samples that can be studied in the future to assess cellular function and fitness for transplant.

Secondary objectives

* To develop gene transfer and gene editing strategies as potentially curative therapy for hemoglobinopathies (e.g. sickle cell disease (SCD) and β-thalassemia).
* To develop a drug treatment strategy which elevates the expression of fetal hemoglobin to a potentially curative level for hemoglobinopathies.
* To examine the biology of bone marrow cells isolated from patients with hemoglobinopathies.

DETAILED DESCRIPTION:
The hemoglobinopathies (e.g. sickle cell disease (SCD) and thalassemia) are devastating inherited anemias that shorten and reduce quality of life. The only current curative therapy for SCD is bone marrow transplantation. However, many patients lack access to suitable donors for transplant. Alternative treatments based on gene therapy, gene editing and novel drugs are currently being developed and show great promise for hemoglobinopathies. Gene therapy and gene editing are especially appealing because they eliminate both the need for donors and the potentially devastating side effects of Graft-versus-Host Disease because they take advantage of the patients own cells. In gene therapy approaches, hematopoietic stem and progenitor cells (HSPCs) are collected from a patient and then treated to 'correct' or 'replace' the disease-causing mutation. However, much work remains to develop optimal gene therapy and gene editing protocols, as well as better understand the inherent biology of HSPCs in patients with hemoglobinopathies.

Researchers at St. Jude want to learn how to best manipulate HSPCs from hemoglobinopathy patients with gene therapy and gene editing technologies to achieve optimal gene correction and/or replacement, as well as optimal engraftment of 'corrected' HSPCs after transplantation. St. Jude researchers also seek to test candidate drugs on SCD HSPCs that might ameliorate the symptoms of SCD. Finally, St. Jude researchers seek to thoroughly characterize the basic biology and function of HSPCs isolated from hemoglobinopathy patients.

Bone marrow-containing bone samples that are typically discarded during orthopedic surgery will be saved from hemoglobinopathy patients, as well as non- hemoglobinopathy patients, undergoing these surgeries. These samples will be shipped to the St. Jude Hematology Department for experimental research aimed at addressing the primary and secondary objectives of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age receiving orthopedic surgery for clinical management that involve bone marrow containing bone discard.
* Patients receiving orthopedic surgery for clinical management will be considered for this study if they have the following diagnosis and criteria:

  * Homozygous S/S disease or doubly heterozygous for S and β thalassemia who are two years or older are eligible.
  * HbE-β- thalassemia or homozygous (severe) β-thalassemia. including those who are transfusion dependent (major) or severely anemic but relatively transfusion independent (intermedia). Diagnostic criteria include standard hematological parameters, red cell indices, hemoglobin electrophoresis and quantitative determination of HbF and HbA2.

Exclusion Criteria:

* Active, acute manifestations of sickle cell disease including painful crisis, acute chest syndrome, cerebrovascular events or active infection.
* Pregnant women will not be eligible for study enrollment
* Inability or unwillingness of the research participant or legal guardian/representative to give written informed consent will preclude enrollment on this research protocol.
* Platelet count < 150,000/mm^3
* Neutrophil count < 2000/mm^3
* Neutrophil count < 1000/mm^3 for patients on hydroxyurea therapy
* Prothrombin Time > 17 seconds
* Partial thromboplastin Time > 43 seconds
* History of excessive bleeding in the context of previous procedures including surgery and dental extractions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who meet the Eligibility Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Collection, processing and storage of discarded bone marrow-containing bone samples from hemoglobinopathy, as well as non-hemoglobinopathy individuals. | After completion of sample collection, approximately 10 years
  Discarded bone marrow-containing bone samples will be collected for use in research; The processing of samples will help to understand how best to manipulate HSPC's from hemoglobinopathy patients with gene therapy and gene technologies in the laboratory environment. It will also allow us to establish a reservoir of samples that can be studied in the future to assess cellular function and fitness for transplant. Samples may be subject to comprehensive assessment of hematopoietic activity using tissue culture based assays, as well as molecular profiling studies of global transcriptome and epigenomes.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon McKinney-Freeman, Ph.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — https://www.stjude.org
- See also: Clinical Trials Open at St. Jude — https://www.stjude.org/protocols